CLINICAL TRIAL: NCT02293278
Title: Preschoolers Activity Trial - a Pilot Randomized Controlled to Increase Physical Activity and Reduce Sedentary Behaviour
Brief Title: Preschoolers Activity Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy Active Living and Obesity Research Group (Other)
Collaborators: University of Victoria (Other); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 10/85X
Record Dates: First submitted 2014-09-29; First posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
Keywords: MVPA; sedentary behaviour; PA intervention; preschool; gross motor; anthropometrics; day care
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Intervention (Experimental): The intervention consists of 2, 3-hour workshops conducted by a master trainer with experience in promoting PA in preschoolers. Each provider in the intervention group is given the Healthy Opportunities for Preschoolers resource training manual, suggested implementation, and a starter kit of equipment. Master Trainers facilitated biweekly PA sessions throughout the intervention.
  During the 6 month intervention, Preschoolers Activity Trial staff will visit the day care facilities to conduct baseline, 3 month, and 6 month measurements.
  Interventions: Behavioral: Physical Activity Intervention
- Control Group (No Intervention): Day cares randomly assigned to the control group will continue with their existing programming. Day care providers will receive the PA intervention upon completion of their involvement in the 6 month trial, including: 2 three hour educational workshops, Healthy Opportunities for Preschoolers manual and program outlining the ideal implementation of activities from the manual.
  During the 6 month intervention, Preschoolers Activity Trial staff will visit the day care facilities to conduct baseline, 3 month, and 6 month measurements.

INTERVENTIONS:
Behavioral: Physical Activity Intervention — The intervention consists of 2, 3-hour workshops conducted by a master trainer with experience in promoting PA in preschoolers. The workshops focus on the importance of PA and movement skills for preschool-aged children, understanding structured and unstructured play, practical activities related to movement skills, how to overcome barriers in facilitating PA, and using everyday materials to facilitate PA and active play. Each provider in the intervention group is given the Healthy Opportunities for Preschoolers resource training manual, suggested implementation, and a starter kit of equipment. Master Trainers facilitated biweekly PA sessions throughout the intervention. The intervention is based on NASPE (2002) guidelines of not having children sedentary more than 60 mins at a time, having children accumulate 60 mins in structured and unstructured PA (active play) each day at MVPA, as well as 180 mins of total PA as recommended by the Canadian PA Guidelines for preschoolers.
  Arms: Physical Activity Intervention

SUMMARY:
The purpose of this pilot study is to test the efficacy of the physical activity (PA) intervention protocol to increase preschoolers overall PA levels and time spent in moderate to vigorous PA (MVPA) at the day care setting. The PA intervention includes the Healthy Opportunities for Preschoolers manual, a compilation of locomotor, gross motor and movement based activities developed for preschoolers and successfully piloted for feasibility in 3 to 5 year old preschoolers by Drs. Viviene Temple, Justen O'Connor, and Patti-Jean Naylor. As well, the PA intervention includes educational workshops for the day care providers, ongoing biweekly facilitation and troubleshooting sessions with a Master Trainer, and the equipment necessary to implement the program. The study is also evaluating the efficacy of the PA intervention to decrease the amount of time spent in sedentary behaviour at the day care setting.

Secondary objectives include evaluating the effects of the PA intervention on preschool children's anthropometrics, and fundamental and gross motor skills. In addition, the intervention is also assessing the effects of the program on day care provider's attitudes, control beliefs, and self-efficacy toward incorporating PA into the day care curriculum.

DETAILED DESCRIPTION:
Background & Significance:

Objective measures of physical activity (PA) using accelerometers (motion sensors worn at the hip) reveal that preschoolers level of sedentary behaviour are high, and levels of moderate to vigorous physical activity (MVPA) are low (Pate et al., 2004, Reilly et al., 2004, 2006). Inquiry into preschoolers daily levels of PA suggest that 2.6% to 4% of waking hours are spent in MVPA (Reilly, 2004, 2006;Montgomery et al. 2004), and, during pre-school hours, Pate and colleagues found that 3 to 5 year old children engaged in 7.7 minutes of MVPA. A recent study of Canadian preschoolers found remarkably similar levels of MVPA (Temple et al., 2009), that include 12.3 minutes of MVPA per day and 39.5 minutes of sedentary behaviour per hour. Although Pate et al. 2004 found that boys had higher levels of MVPA than girls, they did not detect differences in levels of sedentary behaviour, which constituted the vast majority of time for boys and girls. The findings suggest that young children are very inactive and therefore may be at risk for adverse health consequences related to physical inactivity.

Opportunities for PA and motor development in early childhood may, over the lifespan, influence health behaviours and the potential to maintain a healthy body weight. Fundamental movement skills (e.g., catching, throwing, jumping, running, etc.) are the essential building blocks for the acquisition of more refined and complicated skills that can be applied later in life, such as sporting, recreational and physical activities (Gallahue et al. 2002; Carson 1994; Seefeldt, 1979). However, movement skills will not develop to their potential without opportunities to practice in environments that are stimulating and supportive (Kelly et al., 1989; Taggart & Keegan, 1997). Butcher & Eaton found that preschoolers movement competence already influenced their PA choices and levels. It is the mastery of motor skills and the ability of children to incorporate these skills into games, dances, and sports of one's culture that provides the stimulus for movement which contributes to long-term health (Seefeldt & Vogel, 1987).

There is a paucity of information on current trends in PA of preschool aged children, and on the relationship between the ability of children to perform fundamental movement skills and prediction of PA (Mackenzie et al 2003). The few studies noted above indicate that preschool aged children do not come close to being physically active enough to accrue health benefits. In fact, although the evidence of how much and what type of PA is necessary to optimize health and development of preschool-aged children is somewhat unclear (Timmons et al., 2007), expert consensus suggests that preschool-aged children should not be sedentary for more than 60 minutes at a time, except when sleeping, and they should engage in at least 60 minutes (and up to several hours) of structured (facilitated by day care providers, parents, etc. ) and 60 minutes of unstructured PA daily, as well as 180 mins of total PA (National Association for Sport & Physical Education, NASPE, 2002).

In keeping with the settings-based approach to health promotion, which acknowledges the influence of place on behaviour (Dooris et al. 2007), it is believed that powerful influences on children's PA levels are the social and physical environments in which they spend time (Bower et al., 2008; Dowda et al., 2004; Finn eta l., 2002). Over half of all Canadian children aged 6 months to 5 years were in some form of nonparental/guardian care in 2002-2003, and children spent an average of 29 hours a week in these day care settings (Bushnik , 2006; Silver 2000). The majority of Canadian children in both two parent and single parent families fall into this category as 77% of two parent families and 75% of single parent families rely on day care for their children. As such, the paid child day care setting provides an ideal opportunity to examine and enhance the movement skills and PA behaviours of preschool-aged children. There is a small body of evidence that suggests that group preschool and child care settings, policies and practices strongly influence children's PA (Finn et al., 2002; Pate et al., 2004; Bower et al., 2008), but the efficacy of interventions in day care centre settings on preschool children's PA and inactivity behaviours has not yet been determined.

The current PA intervention program is based upon the Healthy Opportunities for Preschoolers manual and program which were developed and successfully piloted for feasibility in 3 to 5 year old preschoolers by Drs. Viviene Temple, Justen O'Connor, and Patti-Jean Naylor. Drs Temple and Naylor are researchers from the University of Victoria, and are co-investigators on this study (Temple et al., 2009). We are using a randomized controlled trial design to build on their previous work to evaluate the efficacy of the physical activity intervention training manual and program to increase PA (with slight modifications and editing of the Healthy Opportunities for Preschoolers training manual).

The Preschoolers Activity Trial was developed from a socio-ecological perspective recognizing that behaviour is affected by multiple levels of influence: intrapersonal, interpersonal, organizational/environmental, community and policy levels. (Burkman & Kawachi, 2000). The program is an environmentally-based intervention and focuses on child care as a setting of influence in children's lives. Recent research has demonstrated the potential of focusing on settings to modify health promoting behaviours such as eating, PA and tobacco use (Snyder et al., 1992; Moore et al., 2001; McKenzie et al., 1994) Theoretically, the focus on the setting is underpinned by the work of community psychologists Barker (1968) and Bronfenbrenner (1999). Behaviour settings are stable units that affect more than one individual and substantially influence the behaviour that occurs within them (Barker, 1968). Barker's research showed that some attributes varied less across children within settings than between settings. Bronfenbrenner's (1999) bio-ecological model expanded this, highlighting the importance of reciprocal interactions in children's development; and the need for children to engage in activities regularly over extended periods of time.

Ultimately, the effectiveness of the PA intervention will rest in our ability to transfer knowledge to the day care-providers which would motivate them to change the child care programming and environment in which children spend time. Despite varying definitions, the measure of effective knowledge transfer or exchange is knowledge utilization (Cousins & Leithwood, 1993); the uptake and implementation of innovation to the curriculum (evidence-based practices) by decision-makers and practitioners.

Study Design and Methodology:

A Cluster randomized controlled trial design will be used with day care centres as the unit of measurement (clusters), though analysis will also be at the individual subjects level given the few number of day cares targeted in this study. Several large (non-home based) day care centres in Ottawa that represent ethnic diversity and varying levels of socio-economic status (SES) have been invited to participate. We sent out a letter to a few daycares that expressed interest, outlining the objectives and procedures of the project, as well as the chance of being randomly assigned to either Intervention or Control Group. The current intervention is designed for 3-5 year old children attending day care. Of the interested day care centres, 3 have been randomly assigned to intervention and 3 to the control group. Day care providers in centres randomized to the control group will receive the educational workshops and the resource manual after their involvement with the study is completed (6 months post-treatment), however the children in the control day care centres will not be evaluated after the providers receive the training.

The PA intervention designed to increase PA and reduce sedentary behaviour consists of 2, three-hour workshop training sessions conducted by a master trainer with experience in promoting PA in preschoolers. The training workshops target the day care providers of 3 to 5 year old children assigned to the intervention group. The first workshop focuses on the importance of PA and movement skills for pre-school-aged children, understanding structured and unstructured play, how to implement HOP in day care centres, and practical activities related to movement skills. The second workshop focuses on overcoming barriers to facilitating PA; understanding the range of movement skills; and using everyday materials to facilitate PA and active play. Each provider in the intervention group is provided with the Healthy Opportunities for Preschoolers resource training manual, a recommended program outlining which activities to participate in and how often, and a starter kit of equipment that forms the basis of training for the day care providers and the intervention. The manual is full of various ways providers can get children active in structured and unstructured physical activities, some of which target motor skill development. The aim of the intervention is based on the aforementioned NASPE (2002) guidelines of not having children sedentary more than 60 minutes at a time, and that children accumulate at least 60 minutes in structured PA and at least 60 minutes of unstructured (active play) each day at moderate intensity or higher.

Participation and Consent:

The parents of children aged 3-5 years, in participating day cares, were given informed consent forms to take home to read. The letter made it clear that the care provider's participation was not dependent on all of the children participating and that their participation was completely voluntary. Participating children receive a randomized identification number, which is used for all data collection, as the information is confidential. This information is linked to a master sheet that is locked in a secure location. Data is collected solely on children who have parental consent.

Questionnaire data:

Day care providers in both groups will be surveyed about their understanding of the Central Health Messages (CHM) associated with Healthy Opportunities for Preschoolers manual, as well as physical facilities in the day care environments that may promote or restrict PA. The questionnaire also assesses providers attitudes, control beliefs, intentions, and support for PA based on the Theory of Planned Behaviour (TPB). Providers will complete these questionnaires at baseline and after the 2 training workshops. This information can then be used to evaluate how well it predicts changes in children's PA and sedentary behaviour. This questionnaire was specifically developed and successfully used in the feasibility and collection of preliminary outcome data in the HOP trial conducted by Drs. Temple and Naylor (co-investigators).

Parents of participating children are sent a socio-demographics questionnaire asking details on parent's age, sex, highest level of education achieved, total parental/family income, height and weight.

Anthropometry and Body Composition Data is collected at each measurement period (baseline, 3 months and 6 months post-intervention workshops):

* Height
* Body weight
* Body mass index (kg/m2)(calculated)
* Body composition (lean body mass, fat mass, and percent body fat) using Bioelctrical impedance analysis validated for the preschool population.

Physical Activity: Self-reported or care provided reports of PA are fraught with difficulties and subject to considerable bias in young children (Adamo et al. 2008). Thus, we are measuring PA objectively using the Actical (mini Mitter Co., Inc., Bend, Ore.) accelerometer which is a small unobtrusive device worn on the right hip by using belts around the waist (in young children), and is an omni-directional sensor to monitor the occurrence and intensity of motion. At each measurement period (baseline, 3- and 6- months post workshop intervention), children wear these activity monitors from the time of awakening (except showering/bathing as they are not waterproof) until the time they go to bed from Monday to Friday, thus providing each subject with a minimum of 4 days of PA monitoring. Parents keep a log to verify times when accelerometers were on and taken off, and whether children napped. To account for the possibility that not all children will wear the Acticals every day, and the length of time that children spend in day care differs, the proportion of PA and sedentary behaviour per hour of wear time will be computed, as done previously in a group of preschool children (Temple et al. 2009). Pfeiffer et al's (2006) cut points for preschool-aged children's moderate and vigorous (MVPA) will be applied. The cut-points will be 715 counts with a 15 second epoch sampling for MVPA,1411 counts using the same 15 second epoch sampling for vigorous PA, and less than 50 counts per hour for sedentary behaviour using a 15 second epoch sampling. For ease of comprehension and comparison with other studies, activity data will be summarized and reported as activity minutes per hour, computed from tallied counts for each activity level average across wear time. Only children with 4 or more hours of accelerometer data per day will be included in the dataset. Acticals will be used to assess overall levels of PA, PA intensity, and energy expenditure at baseline, 3- and 6- months post-intervention.

Fundamental/Gross Motor Skills: We are using the Test of Gross Motor Development -2 (TGMD-2) to evaluate the effects of the intervention on children's movement skills (Ulrich, 2000). The TGMD-2 is a validated standardized norm-referenced measure of 12 common gross motor skills of children ages 3 to 11 years (Evaggelinou et al., 2002). Reliability of the Gross Motor composite index in our targeted age range of children is 0.91 (Ulrich, 2000). Since this test takes about 30-40 minutes, it is conducted on a sub-group (about 50%) of children in both groups to provide pilot data on trends in motor skill development that can inform a larger and more definitive RCT test of HOP. Children in each group are randomly selected to do the TGMD-2 at each measurement time period (baseline, 3- months and 6-months).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 3 to 5 years old
* Enrolled full-time at a participating, licensed daycare/child care facility

Exclusion Criteria:

* Activity restrictions due to disease: unstable cardiac or pulmonary disease, significant arthritis
* Other illness judged by the parent/guardian to make participation in this study inadvisable
* Significant cognitive deficit resulting in inability to understand or comply with instructions
* Inability to communicate in English or French
* Unwillingness of parent/guardian to sign informed consent

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Increase MVPA | 6 months
  Moderate to vigorous physical activity (MVPA) is measured objectively with the children wearing Actical accelerometers for one week. MVPA measured in minutes per day.

SECONDARY OUTCOMES:
Effect of PA intervention on anthropometrics of preschoolers. | 6 months
  Anthropometrics measured include height in metres (using stadiometer), weight in kg (using medical grade scale), body mass index calculated in kg/m2, lean body mass in kg, fat mass in kg, and percent body fat (using bio-electrical impedance)
Effect of PA intervention on fundamental and gross motor skills of preschoolers. | 6 months
  To evaluate the effects of PA intervention on fundamental and gross motor skills in preschoolers attending day care. Gross motor skills will evaluated utilizing the Test of Gross Motor Development- 2 (TGMD-2). Gross motor quotient (GMQ) data will be reported.
Effects of PA intervention on day care provider's attitudes, control beliefs and self efficacy. | 6 months
  A questionnaire is completed assessing the effects of PA intervention on day care providers attitudes, control beliefs, and self-efficacy toward incorporating PA into the day care curriculum. Data will be self-reported by daycare providers using a questionnaire developed specifically for the study by the investigators.
Decrease sedentary behaviour | 6 months
  Sedentary behaviour is measured objectively with the children wearing Actical accelerometers for one week. Sedentary behaviour is measured in minutes per day.
Increase Total Physical Activity | 6 months
  Total Physical Activity (TPA) is measured objectively with the children wearing Actical accelerometers for one week. TPA measured in minutes per day and accelerometer counts per day.

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Goldfield, PhD, Principal Investigator — HALO, CHEO RI; Kristi B Adamo, PhD, Principal Investigator — HALO, CHEO RI
Locations (1):
- Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Goldfield GS, Harvey ALJ, Grattan KP, Temple V, Naylor PJ, Alberga AS, Ferraro ZM, Wilson S, Cameron JD, Barrowman N, Adamo KB. Effects of Child Care Intervention on Physical Activity and Body Composition. Am J Prev Med. 2016 Aug;51(2):225-231. doi: 10.1016/j.amepre.2016.03.024. Epub 2016 May 11. PMID 27180030